CLINICAL TRIAL: NCT05908227
Title: Effects of Flow Magnitude on Cardiorespiratory Stability During Nasal High Flow Therapy in Preterm Infants (MASTER Trial)
Brief Title: Effects of Flow Magnitude on Cardiorespiratory Stability During Nasal High Flow Therapy in Preterm Infants
Acronym: MASTER
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2022-02287
Record Dates: First submitted 2023-05-30; First posted 2023-06-18 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Respiratory Distress Syndrome
Keywords: Nasal high flow therapy; Continuous positive airway pressure
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Masking Description: Due to the nature of the study design masking is not possible.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- NHF high (Experimental): Nasal high flow therapy 8L/min
  Interventions: Other: NHF high
- NHF low (Experimental): Nasal high flow therapy 6L/min
  Interventions: Other: NHF low
- NCPAP (Active Comparator): Nasal continuous positive airway pressure 6 cm H20
  Interventions: Other: NCPAP

INTERVENTIONS:
Other: NHF high — Nasal high flow therapy 8L/min.
  Arms: NHF high
Other: NHF low — Nasal high flow therapy 6L/min.
  Arms: NHF low
Other: NCPAP — Nasal continuous positive airway pressure 6 cm H20
  Arms: NCPAP

SUMMARY:
Premature babies often need help breathing for a longer period of time. Traditionally, this is done with a breathing aid called NCPAP (nasal continuous positive airway pressure). This treatment is safe and effective, but it is very time-consuming and can sometimes have side effects. In the present research project, the investigators want to find out whether another type of breathing aid called NHF (nasal high flow therapy) is just as effective for stable premature babies. The investigators suspect that NHF is just as effective, but easier to use and more comfortable.

DETAILED DESCRIPTION:
This is a multi center parallel group three arm randomized controlled clinical trial investigating cardiorespiratory stability in stable preterm infants receiving NHF.

Currently, NCPAP remains the gold standard for administration of prolonged non-invasive ventilatory support in very preterm infants. NHF is a promising method for tailored, less invasive long-term ventilatory support for preterm infants. If ventilatory support with NHF is similarly effective to conventional NCPAP in stable preterm infants, clinicians are likely to adopt this method for widespread clinical use because of its improved comfort and potential other benefits. Primary aim of this trial is to examine cardiorespiratory stability in preterm infants treated with two commonly used NHF flowrates (Interventional group 1 and 2) in comparison to NCPAP (Comparator). Secondary aim is to examine potential comfort-related beneficial effects of NHF.

ELIGIBILITY:
Inclusion Criteria:

Inclusion if all apply.

* Preterm infants up to 31+6 weeks GA admitted to the Division of Neonatology at Inselspital Bern, Switzerland or Division of Neonatology at the University Medical Center of the Johannes Gutenberg-University Mainz, Germany (inborn or outborn)
* >2nd day of life (defined as date day)
* Stable on NCPAP 6 cm H2O for ≥ 24 hours, defined as:

  * ≤ 2 apneas with concomitant bradycardias (<100/min) per hour for the previous 6 hours
  * FiO2 ≤ 0.3 and not increasing
  * No significant chest recessions (Silverman Score < 5)
  * Respiratory rate ≤ 60/min
  * No need for intermittent positive pressure ventilation
* Parents with an age 18+ years
* Written parental informed consent (or other legal representative)

Exclusion Criteria:

Exclusion if any applies.

* Significant fetal anomalies
* Primary palliative care
* Stable on NCPAP 6 cm H2O according to stability criteria for more than 120 hours

Ages: 23 Weeks to 31 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Treatment failure | 24 hours
  Treatment failure is a composite outcome defined as meeting one of the following treatment failure criteria within 24 hours of starting of intervention:
  1. >2 apneas with concomitant bradycardias (<100/min) per hour for > 1 hour or
  2. FiO2 > 0.3 consistently for > 1 hour or
  3. Significant chest recessions (Silverman Score ≥ 5) for > 1 hour or
  4. Respiratory rate > 60/min consistently for > 1 hour or
  5. Any need for intermittent positive pressure ventilation
  The presence of "Treatment failure" within 24 hours of starting of intervention will be documented (dichotomous outcome; yes/no).

SECONDARY OUTCOMES:
Apneas and bradycardias | 24 hours
  The total frequency of apneas and bradycardias (<100/min) within 24 hours of starting of intervention will be documented.
Respiratory rate (RR) | 24 hours
  The mean RR within 24 hours of starting of intervention will be documented.
Heart rate (HR) | 24 hours
  The mean HR within 24 hours of starting of intervention will be documented.
Oxygen saturation (SpO2) and fraction of inspired oxygen (FiO2) | 24 hours
  The mean SpO2/FiO2 ratio within 24 hours of starting of intervention will be documented.
Frequency of any treatment failure | Individual study duration: estimated to be between a minimum of 7 days to an (estimated) maximum of 10 weeks.
  Treatment failure is a composite outcome (see "Outcome 1"). The frequency of any treatment failure during the duration of the study will be documented.
Rescue NCPAP | Individual study duration: estimated to be between 7 days to 10 weeks.
  Rescue NCPAP is defined as NCPAP >6 cm H2O. The frequency of need for Rescue NCPAP during the duration of the study will be collected.
Postmenstrual age (PMA) off positive pressure support | Estimated to be at a PMA of approximately 29 to 34 weeks.
  The investigators will document the PMA when the infant is off positive pressure support.
Postmenstrual age (PMA) off FiO2 > 0.21 | Estimated to be at a PMA between approximately 28 to 34 weeks.
  The investigators will document the PMA when the infant is off FiO2 > 0.21
Postmenstrual age (PMA) at discharge | Estimated to be at a PMA of approximately 38-40 weeks.
  The investigators will document the PMA when the infant is being discharged from the hospital.
Cerebral oxygen saturation (cRSO2) 1 hour before until 3 hours after start of the intervention | 4 hours
  The cerebral oxygen saturation (cRSO2) in [%] 1 hour before until 3 hours after start of the intervention will be measured by using Near-infrared spectroscopy (NIRS).
Time spent <55% cRSO2 1 hour before until 3 hours after start of the intervention | 4 hours
  The time spent <55% cRSO2 in [min] 1 hour before until 3 hours after start of the intervention will be measured by using Near-infrared spectroscopy (NIRS).
Cerebral oxygen saturation (cRSO2) 1 hour before until 3 hours after cessation of the intervention | 4 hours
  The cerebral oxygen saturation (cRSO2) in [%] 1 hour before until 3 hours after cessation of the intervention will be measured by using Near-infrared spectroscopy (NIRS).
Time spent <55% cRSO2 1 hour before until 3 hours after cessation of the intervention | 4 hours
  The time spent <55% cRSO2 in [min] 1 hour before until 3 hours after cessation of the intervention will be measured by using Near-infrared spectroscopy (NIRS).
Change in end-expiratory lung impedance (ΔEELI) | 48 hours
  The change Δ in end-expiratory lung impedance (ΔEELI) will be measured using electrical impedance tomography (EIT) at 9 different timepoints during the first 48 hours after starting of intervention. One measurement will last 6 minutes.
  The measurements will take place:
  * within 30 minutes before starting of intervention (baseline measurement)
  * 3 minutes before until 3 minutes after starting of intervention
  * within 30 minutes after starting of intervention
  * 2, 6, 12, 24, 36, and 48 hours after starting of intervention
Change in global inhomogeneity (ΔGI) index | 48 hours
  The change Δ in global inhomogeneity (ΔGI) index will be measured using electrical impedance tomography (EIT) at 9 different timepoints during the first 48 hours after starting of intervention. One measurement will last 6 minutes.
  The measurements will take place:
  * within 30 minutes before starting of intervention (baseline measurement)
  * 3 minutes before until 3 minutes after starting of intervention
  * within 30 minutes after starting of intervention
  * 2, 6, 12, 24, 36, and 48 hours after starting of intervention
Change in variability of tidal volume (ΔTV) | 48 hours
  The change Δ in variability of tidal volume (ΔTV) will be measured using electrical impedance tomography (EIT) at 9 different timepoints during the first 48 hours after starting of intervention. One measurement will last 6 minutes.
  The measurements will take place:
  * within 30 minutes before starting of intervention (baseline measurement)
  * 3 minutes before until 3 minutes after starting of intervention
  * within 30 minutes after starting of intervention
  * 2, 6, 12, 24, 36, and 48 hours after starting of intervention
Change in ratio of tidal volume anterior/posterior (ΔRatio TV ap) | 48 hours
  The change Δ in ratio of tidal volume anterior/posterior (ΔRatio TV ap) will be measured using electrical impedance tomography (EIT) at 9 different timepoints during the first 48 hours after starting of intervention. One measurement will last 6 minutes.
  The measurements will take place:
  * within 30 minutes before starting of intervention (baseline measurement)
  * 3 minutes before until 3 minutes after starting of intervention
  * within 30 minutes after starting of intervention
  * 2, 6, 12, 24, 36, and 48 hours after starting of intervention
Incidence of Bronchopulmonary dysplasia (BPD) | At 36 weeks PMA
  The incidence with specification of severity of BPD at 36 weeks PMA will be documented. BPD is a form of chronic lung disease (CLD).
  BPD is classified into 3 levels of severity according to the internationally used definition of Jobe and Bancalari (1).
  FiO2 >0.21 for ≥ 28 days and
  1. Breathing room air (mild)
  2. FiO2 <0.3 (moderate)
  3. FiO2 ≥ 0.3 and/or positive pressure support (severe)
  (1) Jobe AH, Bancalari E. Bronchopulmonary dysplasia. Am J Respir Crit Care Med. 2001;163(7):1723-9.
Urinary cortisol | 24 hours
  A 24-hour-urine-sample will be collected on the third study day. The urinary production rates of cortisol and the most important metabolites will be documented as an indicator for infant stress.
COMFORTneo score | 72 hours
  The COMFORTneo score will be documented on the third, fourth and fifth study day. The score measures comfort and chronic pain by observation.
Revised Bernese Pain Scale for Neonates (BSN-R) score | 72 hours
  The BSN-R score will be documented on the third, fourth and fifth study day. The score measures pain.
Parental assessment of comfort | 72 hours
  The parents will be asked 3 predefined questions concerning their infants' comfort on the on the third, fourth and fifth study day.
NASA Task Load Index (NASA-TLX) | 72 hours
  The NASA-TLX will be filled out by the participants' nurses on the third, fourth and fifth study day. The NASA-TLX is a questionnaire that measures workload.
Nasal trauma score | Individual study duration: estimated to be between 7 days to 10 weeks.
  The nasal trauma score is assessed according to internal standard guidelines in case of a present nasal trauma. The highest respective score and time of assessment will be documented on the participant CRF at 36 weeks PMA. Measuring nasal trauma using the Nasal trauma score takes approximately 20 seconds.
Behavioral Sleep stage classification for Preterm Infants (BeSSPI) | 24 hours
  Sleep-wake cycles as determined by the BeSSPI on the fourth study day will be documented. The BeSSPI identifies sleep stages by observation and takes approximately 2.5 hours.
Parental Bonding Questionnaire (PBQ) | At 36 weeks PMA
  The score of the PBQ will be documented at 36 weeks PMA. The PBQ investigates infant-parental bonding.
Age at initiating breastfeeds | Estimated to be between 30-34 weeks PMA.
  The postmenstrual age (PMA) at initiating breastfeeds will be documented. This refers to the PMA at which the first successful breastfeeding attempt takes place.
Age at reaching full breastfeeds | Estimated to be between 34-40 weeks PMA.
  The postmenstrual age (PMA) at reaching full breastfeeds will be documented. This corresponds to 100% nutrition per breastfeeds for 24 consecutive hours.
Weight | At 36 weeks PMA
  The weight in [g] at 36 weeks postmenstrual age (PMA) will be documented.
Head circumference | At 36 weeks PMA
  The head circumference in [cm] at 36 weeks postmenstrual age (PMA) will be documented.

CONTACTS AND LOCATIONS:
Overall Officials: André Kidszun, Prof. Dr. med., Principal Investigator — Division of Neonatology, Department of Pediatrics, Inselspital
Locations (2):
- University Medical Center of the Johannes Gutenberg-University Mainz, Mainz, Rhineland-Palatinate, Germany
- Department of Pediatrics, Inselspital, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Jobe AH, Bancalari E. Bronchopulmonary dysplasia. Am J Respir Crit Care Med. 2001 Jun;163(7):1723-9. doi: 10.1164/ajrccm.163.7.2011060. No abstract available. PMID 11401896